CLINICAL TRIAL: NCT02425137
Title: A Study of S-1 in Combination With Gemcitabine as First-Line Treatment in Patients With Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TTY Biopharm (Industry)
Collaborators: National Cheng-Kung University Hospital (Other); National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTYTG1308
Record Dates: First submitted 2015-03-26; First posted 2015-04-23 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2017-07

CONDITIONS: Advanced Biliary Tract Cancer(BTC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-1/Gemcitabine (Experimental): single-arm
  Interventions: Drug: S-1/Gemcitabine

INTERVENTIONS:
Drug: S-1/Gemcitabine — Eligible patients will receive gemcitabine 800 mg/m2/day on day 1 and S-1 orally 80-120 mg/day (depending on patient's body surface area (BSA)) on day 1 to 10 in a 2-week cycle.
  Other Names: TS-1/Gemmis

SUMMARY:
Primary Objective:

To evaluate disease control rate (DCR) of S-1 in combination with gemcitabine in patients with advanced biliary tract cancer

Secondary Objectives:

* To evaluate overall response rate (ORR)
* To evaluate progression-free survival (PFS)
* To evaluate overall survival (OS)
* To assess the safety profile

ELIGIBILITY:
Inclusion Criteria:

* 1.histologically confirmed biliary tract carcinoma (including intrahepatic bile duct, extrahepatic bile duct, gallbladder, and ampulla of vater);
* 2.metastatic or unresectable disease;
* 3.no history of chemotherapy or radiotherapy for biliary tract cancer;
* 4.presence of at least one measurable tumor lesion which is defined as lesions that can be accurately measured in at least 1 dimension with longest diameter (LD) ≥20 mm using conventional techniques or ≥10 mm with spiral CT and MRI; measurable lymph nodes must be ≥15 mm in the short axis;
* 5.adequate hematopoietic function which is defined as below:

  1. hemoglobin level ≥ 9 g/dL;
  2. absolute neutrophil count (ANC) ≥ 1,500/mm3;
  3. platelet count ≥ 100,000/mm3;
* 6.adequate hepatic function which is defined as below:

  1. total bilirubin ≤ 1.5 times upper limit of normal (ULN) and < 2 mg/dL, or total bilirubin < 3 mg/dL if biliary drainage was performed;
  2. Alanine aminotransferase (ALT) ≤ 3 x ULN or ALT ≤ 5 x ULN in the presence of liver metastasis;
* 7.adequate renal function: creatinine clearance rate (CCr) ≥ 60 mL/min ((based upon 24-hour urine collection or calculated by Cockroft-Gault formula);
* 8.age of 20 years or above;
* 9.ECOG performance status 0-1;
* 10.life expectancy of at least 12 weeks;
* 11.ability to take oral medication;
* 12.ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* 1.other malignancy within the past 5 years except for adequately treated basal or squamous cell skin cancer or cervical cancer in situ;
* 2.history or known presence of brain metastasis;
* 3.presence of grade 2 or above ascites or pleural effusion;
* 4.presence of grade 2 or above diarrhea;
* 5.presence of mental disease or psychotic manifestation;
* 6.active or uncontrolled infection;
* 7.significant medical conditions that is contraindicated to study medication or render patient at high risk from treatment complications based on investigator's discretion;
* 8.pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential. Patients with childbearing potential shall have effective contraception for both the patient and his or her partner during the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 2 years
  Disease control is defined as having confirmed complete or partial response or stable disease

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  To assess Objective response rate (ORR)
progression-free survival (PFS) | 2 years
  To assess progression-free survival (PFS)
overall survival (OS) | 2 years
  To assess overall survival (OS)
safety profile (percentage of patients with at least one occurrence of preferred term will be included,according to the most severe NCI-CTCAE v4.03 grade) | 2 years
  The incidence and percentage of patients with at least one occurrence of preferred term will be included,according to the most severe NCI-CTCAE v4.03 grade

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, M.D., Principal Investigator — National Institute of Cacer Research, National Health Research Institiutes
Locations (4):
- Taiwan (4):
  - Chang Gung Memorial Hospital, Linkou District
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Result] Morizane C, Okusaka T, Mizusawa J, Takashima A, Ueno M, Ikeda M, Hamamoto Y, Ishii H, Boku N, Furuse J. Randomized phase II study of gemcitabine plus S-1 versus S-1 in advanced biliary tract cancer: a Japan Clinical Oncology Group trial (JCOG 0805). Cancer Sci. 2013 Sep;104(9):1211-6. doi: 10.1111/cas.12218. Epub 2013 Jul 25. PMID 23763511
- [Derived] Chiang NJ, Chen MH, Yang SH, Hsu C, Yen CJ, Tsou HH, Su YY, Chen JS, Shan YS, Chen LT. Multicentre, phase II study of gemcitabine and S-1 in patients with advanced biliary tract cancer: TG1308 study. Liver Int. 2020 Oct;40(10):2535-2543. doi: 10.1111/liv.14538. Epub 2020 Jun 9. PMID 32463975
- See also: TFDA — http://www.fda.gov.tw/TC/index.aspx